CLINICAL TRIAL: NCT06777628
Title: Immunophenotype of Peripheral Blood Mononuclear Cells to Early Predict Response to Immunotherapy in Hepatocellular Carcinoma
Brief Title: Immunophenotype of PBMC to Early Predict Response to Immunotherapy in Hepatocellular Carcinoma
Acronym: Immunecheck
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: Immunecheck
Record Dates: First submitted 2024-11-28; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-09

CONDITIONS: Liver Cancer, Adult
Keywords: immunophenotype; HCC patients; immunotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Angiogenesis Inhibitors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — peripheral blood mononuclear cells separated by Ficoll gradient
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HCC patients: Patients with advanced HCC undergoing immunotherapy
  Interventions: Drug: Immunochemotherapy combined with antiangiogenic

INTERVENTIONS:
Drug: Immunochemotherapy combined with antiangiogenic — Immunochemotherapy combined with antiangiogenic

SUMMARY:
The study is aimed to test the performance of a simple, easy, reproducible cytofluorimetric assay to complement imaging studies for:

* predicting response to immune-therapeutic regimens in HCC in the early phase of treatment,
* to rule out pseudo-progression,
* to early predict the escape from effectiveness of treatment.

DETAILED DESCRIPTION:
* To assess the accuracy of biomarkers from an immunophenotypic test (CD8+, PD1+, PD-L1+, CTLA4+, LAG3+, CD8+PD1+, CD8+PDL1+ peripheral lymphocyte populations and circulating granulocytes) in predicting the response to immuno-therapy in patients affected by hepatocellular carcinoma (HCC).
* To compare the transcriptomic signatures of peripheral blood mononuclear cells (PBMC) of responders and non-responders (assessed at the first imaging study).

RNAseq data will be validated by RT-PCR in independent prospective cohorts.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* diagnosis of HCC
* execution of laboratory tests and subsequent treatments and follow-up at our center.
* obtained written informed consent to the study participation

Exclusion Criteria:

* immune-related concomitant diseases
* HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with advanced hepatocellular carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2028-10-15 (Estimated)

PRIMARY OUTCOMES:
To find predictive biomarkers of response to immunotherapy in HCC | at 3 month
  Sensitivity and specificity of CD8+, PD1+, PD-L1+, CTLA4+, LAG3+, TIGIT+, CD8+PD1+, CD8+PDL1+ peripheral lymphocytes and granulocytes for tumor response prediction according to RECIST 1.1 criteria

SECONDARY OUTCOMES:
To compare the transcriptomic signatures of PBMC of responders and non-responders | At 3 months
  Tumor response according to RECIST 1.1 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Laura Gramantieri, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS-Azienda Ospedaliero-Universitaria di Bologna, Bologna, Laura Gramantieri, Italy

IPD SHARING:
Plan to Share IPD: Undecided